CLINICAL TRIAL: NCT03533387
Title: Bioequivalence Study of Two MN-166 (Ibudilast) 50 mg Extended Release Tablet Formulations Compared With MN-166 (Ibudilast) 10mg Capsules in Healthy Volunteers
Brief Title: Study of MN-166 (Ibudilast) Extended Release Tablet Formulations Compared With Capsules in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MediciNova (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MN-166-HDT-001
Record Dates: First submitted 2018-04-18; First posted 2018-05-23 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — ibudilast

STUDY DESIGN:
Intervention Model Description: Subjects will receive the following three treatments in a crossover fashion, administered one week apart:
  * ER1: Single dose (50mg) of ER Prototype 1 (one 50mg ER1 tablet),
  * ER2: Single dose (50mg) of ER Prototype 2 (one 50mg ER2 tablet), and
  * IR: Two doses of intermediate-release capsules (50mg Pinatos® capsules in two divided doses 12 hours apart, i.e., 25mg for each dose).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Extended-release formulation 1 (ER1) (Experimental): 50mg MN-166 tablet. This formulation is intended for once-a-day dosing, hence, the label of extended-release.
  Interventions: Drug: MN-166
- Extended-release formulation 2 (ER2) (Experimental): 50mg MN-166 tablet. This formulation is intended for once-a-day dosing, hence, the label of extended-release.
  Interventions: Drug: MN-166
- Intermediate-release formulation (IR) (Active Comparator): 10mg MN-166 capsule. This formulation is typically given two or three times daily, hence, the label of intermediate-release.
  Interventions: Drug: MN-166

INTERVENTIONS:
Drug: MN-166 — an orally available small molecule drug approved in Japan and Korea for asthma and post-stroke complications and has been prescribed for these indications for more than 25 years
  Other Names: ibudilast; Pinatos® capsule

SUMMARY:
To compare the bioavailability and pharmacokinetic profiles of two different formulations MN-166 50mg, extended release (ER) tablets with MN-166 10mg capsules in a single-dose regimen in healthy volunteers

DETAILED DESCRIPTION:
Part 1:

To compare the bioavailability and pharmacokinetic profiles of two different formulations MN-166 50mg, extended release (ER) tablets with MN-166 10mg capsules in a single-dose regimen in healthy volunteers; and To choose one of the two MN-166 50mg ER tablet formulations for evaluation in Part 2.

Secondary: To determine the safety and tolerability of the two formulations of MN-166 ER tablets in a single-dose regimen in healthy volunteers.

Part 2:

To compare the bioavailability and steady-state pharmacokinetic profile of MN-166 50mg ER tablet with MN-166 10mg capsules in a multiple-dose regimen in healthy volunteers; and

Secondary: To determine the safety and tolerability of MN-166 ER tablets in a multiple-dose regimen in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent.
2. Healthy non-smoking male and female subjects aged 18 to 65 years, inclusive.
3. No clinical abnormalities in laboratory and urine analyses.
4. Normal renal function (GFR > 90mL/min).
5. Liver enzymes should be less than twice the upper limit of normal (ULN).
6. Screening electrocardiogram (ECG) with QT interval adjusted for heart rate within normal limits.
7. Agree to use barrier contraceptive methods during the course of the study (hormonal contraceptive alone is not acceptable).
8. Females of child-bearing potential must have a negative pregnancy test on Study Day 1.

Exclusion Criteria:

1. Known hypersensitivity to Pinatos® or its components.
2. Condition(s) which might affect drug absorption, metabolism or excretion.
3. Untreated mental illness, current drug addiction or abuse or alcoholism.
4. Donated blood in the past 90 days or have poor peripheral venous access.
5. Platelets < l00,000/mm3, history of thrombocytopenia.
6. Confirmed diagnosis of chronic liver disease, e.g., chronic Hep. B, Hep. C infection, auto-immune, alcoholic or neoplastic liver disease.
7. Positive serostatus for HIV.
8. Currently pregnant or nursing.
9. History of clinically significant cardiovascular, pulmonary, endocrine, neurological, metabolic, or psychiatric diseases.
10. Received an investigational drug in the past 30 days.
11. Unable to swallow tablets.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2018-07-06 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Compare the PK Profile of two new formulations in Single-day dose of MN-166 | 5 weeks
  Compare the maximum plasma concentrations [Cmax] of MN-166 of two different formulations MN-166 50mg, extended release (ER) tablets with MN-166 10mg capsules in a single-dose regimen in healthy volunteers.

SECONDARY OUTCOMES:
Compare the incidence of treatment-emergent adverse events of two new formulations in Single-day dose of MN-166 | 5 weeks
  Compare the number and frequency of treatment-emergent adverse events (serious and non-serious) profiles of two different formulations MN-166 50mg, extended release (ER) tablets with MN-166 10mg capsules in a single-dose regimen in healthy volunteers.
Compare the PK Profile of two new formulations in Multi-day dose of MN-166 | 3 weeks
  Compare the maximum plasma concentrations [Cmax] of MN-166 of two different formula in a multiple-dose regimen.
Compare the incidence of treatment-emergent adverse events of two new formulations in Multi-day dose of MN-166 | 3 weeks
  Compare the number and frequency of treatment-emergent adverse events (serious and non-serious) of MN-166 (pharmacokinetic profiles) of two different formula in a multiple-dose regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Robina Smith, MD, Principal Investigator — WCCT Global, Inc.
Locations (1):
- WCCT Global, Inc., Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No